CLINICAL TRIAL: NCT03497507
Title: Effect of P6 Acupressure Stimulation on Shivering During Cesarean Section Under Epidural Anesthesia.
Brief Title: Investigating the Effect of Acupressure on Shivering During a Cesarean Delivery in Women Who Were Previously Laboring With an Epidural
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Anesthesiologist, Associate professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 17-2495
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Shivering; Labor; Cesarean Delivery
Keywords: Shivering; Cesarean delivery; acupressure; P6 acupoint

STUDY DESIGN:
Intervention Model Description: Once an obstetrician determines that a patient laboring with an epidural catheter should have a non-emergent cesarean section instead of continuing labor, the clinical anesthesiologist will contact the research team. A member of the research team will contact the patient while she is still in the labor and delivery room, at which time informed consent would be obtained.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham bracelet (Placebo Comparator): Patients randomized to sham group will wear bracelets on both hands which will not apply acupressure
  Interventions: Device: Sham bracelet
- Acupressure bracelet (Experimental): Patients randomized to the experimental group will wear bracelets on both hands which will apply acupressure to the P6 acupoint.
  Interventions: Device: Acupressure bracelet

INTERVENTIONS:
Device: Sham bracelet — Patients will wear bracelets on both hands
  Arms: Sham bracelet
Device: Acupressure bracelet — Patients will wear bracelets on both hands.
  Arms: Acupressure bracelet

SUMMARY:
Shivering during a cesarean section can be quite uncomfortable for the patient as well as make it difficult for the anesthesiologist to obtain vital signs. The researchers will investigate whether or not applying pressure to the P6 acupressure point during a cesarean section can treat shivering. The hypothesis is that shivering will be alleviated with acupressure.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether applying pressure to the left and right P6 acupoints can treat shivering in a patient undergoing a cesarean section. The hypothesis is that bilateral stimulation of P6 with pressure can stop or alleviate shivering.

The primary endpoint is resolution of shivering within 15 minutes of applying bilateral pressure to P6 acupoints during a cesarean section.

The secondary endpoints include:

1. Time to resolution of shivering
2. Degree of patient-reported improvement in shivering
3. Degree of practitioner-reported improvement in shivering
4. Assessment of skin irritation and/or pain at the site of acupressure vs control

Patient information will be stored in a locked cabinet on labor and delivery, and that cabinet will be located in a T3-locked office. The link between subject ID and patient ID will be stored in a different office on labor and delivery, also under a T3 lock.

Patients who are laboring with an epidural catheter and subsequently require a cesarean section will be selected. This patient population has a MUCH higher rate of shivering during the cesarean section as compared to patients who undergo elective scheduled cesarean sections under spinal anesthesia. By selecting this group, the investigators are not only increasing chances of identifying shivering but also decreasing variability between patient characteristics by limiting it to one type (only epidural and not spinal) and limiting the number of screen failures.

ELIGIBILITY:
Inclusion Criteria:

* a patient has to be classified as an American Society of Anesthesiology (ASA) physical status I, II, or III, laboring with an epidural catheter, and subsequently taken for a non-emergent cesarean section under epidural anesthesia with a core body temperature range of 35.5-38.0 degrees Celsius during shivering.

Exclusion Criteria:

* ASA status 4 or higher
* core body temperature lower than 35.5 or higher than 38.0
* thyroid disease
* systemic infection
* emergent cesarean section,
* a psychiatric, cognitive or medical condition that would compromise adherence to the protocol

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is studying shivering during a cesarean delivery.
Enrollment: 43 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of resolution of shivering at 15 minutes | up to 15 minutes
  Incidence of resolution of shivering within 15 minutes of applying bilateral pressure to P6 acupoints during a cesarean section.

SECONDARY OUTCOMES:
Time to resolution of shivering | up to 15 minutes
  Time to resolution of shivering
Degree of resolution of shivering | up to 15 minutes
  Degree of patient-reported improvement in shivering as measured by Crossley & Mahajan shivering scale: 0 = no shivering;1 = no visible muscle activity but piloerection, peripheral vasoconstriction, or both are present (other causes excluded); 2 = muscular activity in only one muscle group; 3 = moderate muscular activity in more than one muscle group but no generalized shaking; 4 = violent muscular activity that involves the whole body.
Degree of practitioner-reported improvement in shivering | up to 15 minutes
  Degree of practitioner-reported improvement in shivering as measured by Crossley & Mahajan shivering scale: 0 = no shivering;1 = no visible muscle activity but piloerection, peripheral vasoconstriction, or both are present (other causes excluded); 2 = muscular activity in only one muscle group; 3 = moderate muscular activity in more than one muscle group but no generalized shaking; 4 = violent muscular activity that involves the whole body.
Number of participants with skin irritation | up to 15 minutes
  Number of participants with skin irritation at the site of acupressure obtained by patient self-reporting
Number of participants with pain | up to 15 minutes
  Number of participants with pain at the site of acupressure obtained by patient self-reporting

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Zahn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided